CLINICAL TRIAL: NCT00164060
Title: Associations, Outcomes and Genomics of GB Virus C, Hepatitis C Virus and Human Immunodeficiency Virus Infection
Status: Terminated | Type: Observational
Sponsor: Bayside Health (Other Government)
Other Study IDs: 35/04
Record Dates: First submitted 2005-09-13; First posted 2005-09-14 (Estimated); Last update posted 2013-12-05 (Estimated); Status verified 2005-09

CONDITIONS: Hepatitis C; HIV Infections
Keywords: HCV; HIV co-infection
MeSH Terms: conditions — Hepatitis C; HIV Infections

STUDY DESIGN:
Time Perspective: Retrospective

SUMMARY:
The purpose of this study is to examine the effect of GB virus C (GBV-C) on the natural history of chronic hepatitis C virus (HCV) infection in subjects co-infected with HIV and HCV. The other aspect of the study is to assess the effect of GBV-C on the severity of liver disease due to chronic hepatitis C in subjects co-infected with HIV and HCV. This will be done by determining the point prevalence of co-infection retrospectively then following that cohort prospectively. In addition, further individuals will be recruited in a prospective manner.

DETAILED DESCRIPTION:
Background and Research Plan:

GBV-C and hepatitis G virus (HGV) are both RNA viruses from the Flaviviridae family. Molecular characterization of these viruses has shown them to be virtually identical to each other (1,2). GBV-C was first isolated in 1995 from an archival blood sample obtained in the 1960s from a surgeon with acute non A-E hepatitis (3). GBV-C has a 29% amino acid sequence homology with Hepatitis C Virus (HCV), another flavivirus (4). However, GBV-C in contrast to HCV, is not hepatotropic as the virus neither replicates primarily in hepatocytes nor causes acute or chronic hepatitis. Indeed, GBV-C does not cause any specific disease nor does it represent a substantial health risk in humans. Nevertheless, GBV-C infection is relatively common with a 2% prevalence rate in healthy blood donors, the majority of whom clear the virus and develop antibodies to the envelope glycoprotein E2.

HIV infection has a particularly high rate of co-infection with GBV-C. Studies suggest that co-infection leads to a beneficial effect on the course of HIV (5,6,7) with co-infection associated with a significantly lower mortality rate among HIV-infected subjects compared to those not infected with GBV-C. The mechanism of the beneficial effect of GBV-C on the course of HIV infection is obscure.

Among new cases of non-A, non-B hepatitis in the United States, 18 percent are positive for GBV-C, and 80% of these patients are also infected with HCV. Amongst patients with HCV, 10-20% have GBV-C RNA in their serum (4). In another report 189 patients with chronic HCV infection were evaluated; 21 (11%) were positive for GBV-C RNA (8). The course of the HCV infection and the response to interferon-alfa were not affected by co-infection with GBV-C. Interferon-alfa led to a decrease in GBV-C RNA titers that was not sustained after the cessation of therapy. Similar findings were noted in another study in which liver biopsies were performed (9). Detailed histopathologic examination revealed no difference between the patients infected with HCV alone and the 15 percent who were co-infected with GBV-C. There have been no studies to date looking at the effect GBV-C, HCV and HIV have on each other.

Our previous studies into HIV and GBV-C have suggested that co-infection is common. Active GBV-C infection is frequently observed in persons involved in high-risk sexual activity and with HIV infection. Homosexual intercourse appears to be a more effective means of transmission of GBV-C. GBV-C has the same epidemiology and transmission as HIV and underlines the intimate association between GBV-C and HIV (10).

Methods/Experimental Design:

Stored sera is available from people who have attended the Hepatitis and HIV clinics at the Alfred Hospital. Sera is available back to approximately 1990 and has been stored at minus 20ºC and as such is suitable for GBV-C detection particularly RNA by PCR. Of the sera stored by the HIV clinic 203 patients are known to be co-infected with HCV who are currently still alive. Once ethics committee approval is obtained we propose to contact these groups of people and see if they would participate in this study. Once consent is obtained we plan to perform the following.

A. Stored sera will be retrospectively examined for the point prevalence of infection with HCV, GBV-C and HIV. These individuals will then be followed up in a prospective manner assessing the progression of liver disease and other factors as outlined in Tables 1 to 4.

B. New subjects attending the Alfred Hospital Hepatitis or HIV clinics will be recruited and followed prospectively also as outlined in Tables 1 to 4.

C. An age and sex matched control group infected with HCV alone will be identified via the Alfred Hospital Hepatitis clinic. This clinic has a large cohort of well-characterized HCV infected subjects that extends back to 1989.

The inclusion and exclusion criteria for the study are as follows:

Inclusion criteria

1. Sera available and appropriate for testing. Including serial sera over a period of time. (retrospective analysis)
2. HIV serology positive.
3. Unequivocal HCV antibody positive or HCV RNA positive.

Exclusion criteria

1. Those without sera available.
2. Those unwilling to give informed consent.
3. Persons with Hepatitis B Virus infection, as defined by the presence of Hepatitis B surface antigen and/or Hepatitis B Virus DNA positive.

Where possible information will also be obtained about these people by interview, examining the medical records or discussion with their General Practitioners. Subjects will also be encouraged to attend the hospital in person where a clinical exam can be performed. If insufficient sera is stored further blood will be drawn at this time and examined for HCV, HIV and GBV-C related parameters as outlined in the tables below. A study specific questionnaire will be generated in which subjects will be asked to complete a confidential questionnaire that contains information related to demographic and behavioral factors that may contribute to the acquisition of GBV-C, HCV or HIV infection or various combinations of the above. Demographic variables will include age, sex, country of birth, and occupation. Information relevant to HIV infection including the use of HAART and the presence or absence of AIDS defining syndromes will be obtained. The questionnaire will attempt to identify the approximate time of acquisition of both HCV and HIV. In addition, the extent of liver disease will be assessed, alcohol consumption will be quantified and information will be gathered on previous treatment with Interferon and Ribavirin.

The main outcomes of this study will be liver related morbidity, such as chronic hepatitis, cirrhosis or hepatocellular cancer and overall patient survival. The detailed information contained in the following tables will be obtained from interview, medical records and clinical examination:

Table 1: GBV-C

1. Testing sera for GBV-C RNA and E2 antibodies to GBV-C.
2. Performing testing at one-year intervals if sera is available.

Table 2: HIV

1. CD4 count (buffy coat) in HIV positive.
2. HIV viral load.
3. Use of highly active antiretroviral therapy (HAART) and other retroviral treatment and/or change in treatment.
4. Complications of HIV/AIDS and AIDS defining illnesses.

Table 3: Liver disease (HCV)

1. HCV viral load and genotype.
2. Child-Pugh classification based on levels of bilirubin, albumin and clotting profiles, and the presence of ascites and encephalopathy.
3. Complications of liver disease: ascites, encephalopathy, variceal bleeding and hepatocellular carcinoma.
4. ALT and AST levels as well as AST/ALT ratio.
5. Alpha Feto Protein (AFP) level.
6. Liver histology at biopsy with assessment of inflammation grade, stage of fibrosis and severity of hepatic steatosis.
7. Liver ultrasound results.
8. Results of endoscopy, i.e. features of portal hypertension

Table 4: Survival Data

1. Has patient died?
2. Date of death.
3. Cause of death.

Results will be statistically examined by univariate and multivariate analysis in terms of clinical outcomes with respect to chronic hepatitis C liver disease between GBV-C positive and negative groups in the HIV co-infected cohort compared with the HCV infected cohort alone. See following Table 5.

Table 5: Study Design

Study Group No.1 HCV +ve, HIV +ve, GBV-C RNA+ve. Study Group No.2 HCV +ve, HIV +ve, GBV-C RNA-ve. Control Group HCV +ve alone.

References relevant to this project (from literature search)

1. Linnen J, Wages J, Zhang-Keck Z, et al. Molecular cloning and disease association of hepatitis G virus: A new transfusion transmissible agent. Science 1996; 271:505-8.
2. Alter HJ. The cloning and clinical implications of HGV and HGBV-C. N Engl J Med 1996; 334:1536-7.
3. Simons JN, Leary TP, Dawson GJ, et al. Isolation of novel virus-like sequences associated with Human hepatitis. Nat Med 1995;1:564-9.
4. Di Bisceglie AM. Hepatitis G virus infection: A work in progress. Ann Intern Med 1996; 125:772.
5. Tillman HL, Heiken H, Knapik-Botor A, et al. Infection with GB virus C and reduced mortality among HIV-infected patients. N Engl J Med 2001; 345:715-24.
6. Xiang J, Wunschmann S, Diekema DJ, et al. Effect of coinfection with GB virus C on survival among patients with HIV infection. N Engl J Med 2001;345:707-14.
7. Lefrere JJ, Roudot-Thoraval F, Morand-Joubert L, et al. Carriage of GB virus C/hepatitis G virus RNA is associated with a slower immunologic, virologic and clinical progression of human Immunodeficiency virus disease in coinfected persons. J Infect Dis 1999; 179:783-9.
8. Tanaka E, Alter HJ, Nakatsuji Y, et al. Effect of hepatitis G virus infection on chronic hepatitis C. Ann Intern Med 1996;125:740-3.
9. Bralet MP, Roudot-Thoraval F, Pawlotsky JM, et al. Histopathologic impact of GB virus C infection on chronic hepatitis C. Gastroenterology 1997;112:188-92.
10. Berzsenyi MD, Bowden SD, Bailey MJ, et al. Sexual and blood-borne transmission of GB virus C and its association with Human Immunodeficiency Virus. In press.

ELIGIBILITY:
Inclusion Criteria:

1. Sera available and appropriate for testing, including serial sera over a period of time (retrospective analysis)
2. HIV serology positive.
3. Unequivocal HCV antibody positive or HCV RNA positive.

Exclusion Criteria:

1. Those without sera available.
2. Those unwilling to give informed consent.
3. Persons with hepatitis B virus infection, as defined by the presence of hepatitis B surface antigen and/or hepatitis B virus DNA positive.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 158 (Actual)
Dates: Start 2004-02; Primary Completion 2007-05 (Actual); Study Completion 2007-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark D Berzsenyi, MBBS, Principal Investigator — Alfred Hospital/Bayside Health; Stuart R Roberts, MBBS, Study Director — Alfred Hospital/Bayside Health
Locations (1):
- Alfred Hospital, Melbourne, Victoria, Australia

REFERENCES:
- [Result] Berzsenyi MD, Bowden DS, Roberts SK. GB virus C: insights into co-infection. J Clin Virol. 2005 Aug;33(4):257-66. doi: 10.1016/j.jcv.2005.04.002. PMID 15922655
- [Derived] Berzsenyi MD, Bowden DS, Kelly HA, Watson KM, Mijch AM, Hammond RA, Crowe SM, Roberts SK. Reduction in hepatitis C-related liver disease associated with GB virus C in human immunodeficiency virus coinfection. Gastroenterology. 2007 Dec;133(6):1821-30. doi: 10.1053/j.gastro.2007.08.076. Epub 2007 Sep 5. PMID 18054555